CLINICAL TRIAL: NCT02494557
Title: Risk Stratification for Coronary Artery Disease With Type 2 Diabetic Patients
Acronym: CAD-risk
Status: Completed | Type: Observational
Sponsor: Acarix (Industry)
Collaborators: Steno Diabetes Center Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: CAD-risk/2014
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for biobank to be used in potential new studies.
Oversight: Data Monitoring Committee: No

SUMMARY:
Diabetic type 2 patients (DB2) has a higher prevalence of coronary artery disease (CAD) than non-diabetic persons. Presence of CAD results in murmurs arising from the filling of the arteries and can be detected by the CADScor System and can together with biological patient profile indicate the risk of presence of CAD in the patient. In the pilot study 100 asymptomatic DB2-patients examined with CADScor System and biomarkers will be compared with computed tomography (CT) cardiography and single-photon emission computed tomography (SPECT) for assessing if combination of patient profile (gender, age etc) combined with above measures may give rise to new improved risk scoring method for he DB2-patient.

DETAILED DESCRIPTION:
The study is intended as a pilot observational study for evaluation of a new risk scoring method, CADScor System, is relevant for assessment of CAD in the DB2-patient.

The primary end point will be to document that the hypothesis of combining the CADScor System measure with other patient profile data will increase the accuracy of the method for determination of risk of presence of CAD.

The secondary endpoint will be to show that a receiver operating characteristic curve (ROC) of > 80% for correct determination of presence of CAD will be achieved.

The further objective of the study will be to confirm the relevance of performing a large scale study with equivalent objectives.

As controls in the study will be applied CT angiography, CT-calcium and resting and drug induced CT-scintigraphy.

It is assumed that 15-20 of enrolled patients in the study will suffer from CAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from diabetes type 2
* Both sexes
* Patients between 40 and 80 years
* Patients without chest pain at rest and labor
* Patients having a normal electrocardiogram (ECG, i.e. without Q-peaks/ T-peak abnormalities in sinus rhythm)
* Patients having intact skin over sternum

Exclusion Criteria:

* Patients suffering from a heart disease
* Patients already having received heart surgery
* Patients with pacemaker or other implanted electronic device
* Patients suffering from allergy against iodine and iodine containing substances
* Patients with estimated GFR below 50 ml/min/1.73 sqm m
* Patients suffering from adenosine intolerance or known allergic asthma
* Patients not being capable of understanding the patient information of the study
* Patients who are pregnant
* Patients suffering from allergy to adhesives

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic type 2 patient
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Acoustic Cad-score | 1 year
  Comparison of an non-invasive acoustic Cad-score as risk prediction for presence of coronary artery disease with control studies of CT-angiography and resting and drug induced CT scintigraphy

SECONDARY OUTCOMES:
The degree of presence of coronary artery disease (CAD) in Diabetic type 2 patients (DB2) patients | 1 year
  Resting and drug induced perfusion test will be compared to CT Angiography for determining the degree of presence of CAD when including patient parameters characterizing the status and severity of the DB2.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, Professor, Principal Investigator — Steno Diabetes Center, Niels Steensensvej 4, 2840 Gentofte, Denmark
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided